CLINICAL TRIAL: NCT02175823
Title: Health Status Evaluation for Cancer Survivors by Non-intrusive Sensing System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401056RIND
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Cancer
Keywords: Cancer survivors; circadian rhythm; Elderly Patients; frailty
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To improve quality of life of elderly cancer survivors

1. Using physical activity and environmental sensing technology
2. Monitoring physiological indicators of cancer recurrence

   * Analyzing the patient's circadian rhythm, frailty and his/her vital sign.
   * Vital sign includes blood pressure, weight and hrv.
3. Collecting the patient information in real time

   * Giving alarm information to the patient, if any special cases our system found.
   * Giving circadian rhythm report to the patient.
   * Giving healthy report to the patient, collected from his/her vital sign.

ELIGIBILITY:
Inclusion Criteria:

* The clinical pathology and diagnostic imaging to determine the cancer who completed acute treatment, and patients with more than a month recuperating.
* Over 65 years old.
* Proficient in Chinese or Taiwanese.
* Normal cognitive function

Exclusion Criteria:

* No history of cancer
* Over 65 years old.
* Proficient in Chinese or Taiwanese.
* Normal cognitive function

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly cancer survivors
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen Fu, Principal Investigator — Computer Science and Information Engineering
Locations (1):
- National Taiwan University Hospital, Taipei, Da'an Dist, Taiwan